CLINICAL TRIAL: NCT06328283
Title: The Diagnostic Efficacy of Glutamine Synthetaseand BCLAF1in Early Diagosis of GLutamine Synthetase and BCLAF1 in Diagnosis of Hepatocellular in Cirrhotic Patients
Brief Title: The Diagnostic Efficacy of Glutamine Synthetaseand BCLAF1in Early Diagosis of Hepatocellular Carcinoma in Cirrhotic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Safwat Abdelrahman, assisstant lecturer in tropical medicine- sohag university, Sohag University
Other Study IDs: Soh-Med-24-02-01MD
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases group: cirrhotic patients with early hepatocellular carcinoma
  Interventions: Other: measure of Glutamine synthetase and BCLFAF1
- control group: cirrhotic patients with no hepatocellular carcinoma
  Interventions: Other: measure of Glutamine synthetase and BCLFAF1

INTERVENTIONS:
Other: measure of Glutamine synthetase and BCLFAF1 — compare Glutamine synthetase and BCLFAF1 in cases and controls

SUMMARY:
Hepatocellular carcinoma (HCC) is the most prominent kind of liver cancer, accounting for 85% of primary liver malignancies. It is a very aggressive tumor, having a terrible prognosis and poor survival rate HCC is ranked as the sixth most common type of cancer and the third leading cause of cancer-related mortalities world wide.

HCC incidences arise in complications associated with chronic liver disease like cirrhosis, endemic hepatitis B virus (HBV)/hepatitis C virus (HCV) infections, non alcoholic fatty liver disease (NAFLD), and alcohol-related liver disease (Torre, 2015).

ELIGIBILITY:
Inclusion Criteria:

* A total 90 adult patients with liver cirrhosis attending the outpatient clinic or in patient section of the department of tropical medicine and gastroenterology at Sohag University Hospital will be included in the study. Patients will be divided into two groups:

Group I:

The study group will include 45 patients diagnosed with liver cirrhosis with absence of hepatic focal lesion as control group. Cirrhosis will be determined according to clinical , sereological ,radiological findings.

Group II:

The study group will include 45 patient with HCC on top of liver cirrhosis .All causes of liver cirrhosis will be accepted .HCC will be assessed by triphasic CT or MRI or histological validation .In these group we will take patients with liver cirrhosis with early hepatocellular carcinoma that defined as tumors smaller than 3cm and three or fewer in number at stage A according to BCLC staging also sometimes it includes solitary tumors up to 5 cm in size as defined in the Milan criteria. Both very early and early stage tumors are relatively small but both are hyper vascular in arterial phase.

Exclusion Criteria:

1. Non cirrhotic patients.
2. Patients with distant metastasis.
3. Patients aged below18 years.
4. Patients with other malignancy rather than HCC.
5. Patients with late stage of HCC.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: - A total 90 adult patients with liver cirrhosis attending the outpatient clinic or in patient section of the department of tropical medicine and gastroenterology at Sohag University Hospital will be included in the study. Patients will be divided into two groups:
  Group I:
  The study group will include 45 patients diagnosed with liver cirrhosis with absence of hepatic focal lesion
  Group II:
  The study group will include 45 patient with HCC on top of liver cirrhosis .
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
glutamine synthetase | 1 year
  to detect early HCC IN CIRRHOTIC

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Sohagm, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mir IH, Guha S, Behera J, Thirunavukkarasu C. Targeting molecular signal transduction pathways in hepatocellular carcinoma and its implications for cancer therapy. Cell Biol Int. 2021 Nov;45(11):2161-2177. doi: 10.1002/cbin.11670. Epub 2021 Aug 1. PMID 34270844
- [Background] Singh G, Yoshida EM, Rathi S, Marquez V, Kim P, Erb SR, Salh BS. Biomarkers for hepatocellular cancer. World J Hepatol. 2020 Sep 27;12(9):558-573. doi: 10.4254/wjh.v12.i9.558. PMID 33033565
- [Background] Terentiev AA, Moldogazieva NT. Alpha-fetoprotein: a renaissance. Tumour Biol. 2013 Aug;34(4):2075-91. doi: 10.1007/s13277-013-0904-y. Epub 2013 Jun 14. PMID 23765762
- [Background] Wasfy RE, Shams Eldeen AA. Roles of Combined Glypican-3 and Glutamine Synthetase in Differential Diagnosis of Hepatocellular Lesions. Asian Pac J Cancer Prev. 2015;16(11):4769-75. doi: 10.7314/apjcp.2015.16.11.4769. PMID 26107238